CLINICAL TRIAL: NCT06672692
Title: A Multi-Site Clinical Evaluation of the LIAISON NES FLU A/B, RSV & COVID-19 Assay in Symptomatic Patients
Acronym: NES ABCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DiaSorin Molecular LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DSM-PROT-005198
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Influenza a; Influenza B; RSV; COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Masking Description: Participants are not provided investigational results and will only be provided with routine standard of care diagnostics results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blinded, Prospective Arm (Other): Clinical specimens shall be collected prospectively from patients with signs or symptoms of respiratory tract infection. Nasal swab in Copan universal transport media (UTM) 3 milliliters for comparator testing should be collected by a healthcare professional.
  Where subjects are willing and able, up to 40% of nasal swab for the investigational device will be self-collected under the guidance and supervision of a healthcare professional.
  Nasopharyngeal (NPS) specimens (optional) should only be collected by a healthcare professional. All specimens collected from children 13 years or younger should only be collected by a trained healthcare professional. Follow the Centers for Disease Control and Prevention guidelines for collecting NPS swabs, unless otherwise specified by the sponsor.
  Interventions: Diagnostic Test: LIAISON NES FLU A/B, RSV & COVID-19

INTERVENTIONS:
Diagnostic Test: LIAISON NES FLU A/B, RSV & COVID-19 — The LIAISON® NES FLU A/B, RSV & COVID-19 assay used on the LIAISON® NES instrument is a real-time PCR system that enables the direct amplification, detection and differentiation of Flu A viral RNA, Flu B viral RNA RSV viral RNA, and SARS-CoV-2 RNA from dry nasal swabs. Nasal Swabs can be professionally collected by a Healthcare Provider or self-collected by the patient under the supervision of the healthcare provider. The collected nasal swab can then be directly loaded into the cartridge without nucleic acid extraction.

SUMMARY:
The DiaSorin Molecular LIAISON® NES FLU A/B, RSV & COVID-19 real-time polymerase chain reaction (RT-PCR) assay is intended for use on the DiaSorin LIAISON® NES instrument for the in-vitro qualitative detection and differentiation of nucleic acid from influenza A, influenza B, RSV and SARS-CoV-2 virus from dry nasal swabs (NS) from human patients with signs and symptoms during the acute phase of respiratory tract infection in conjunction with clinical and epidemiological risk factors.

The LIAISON® NES FLU A/B, RSV & COVID-19 assay is intended for use as an aid in the differential diagnosis of influenza A, influenza B, RSV and SARS-CoV-2 infection in a professional laboratory setting.

Negative results do not preclude influenza A, influenza B, RSV or SARS-CoV-2, infection and should not be used as the sole basis for patient management decisions. The assay is not intended to detect the presence of the influenza C virus.

ELIGIBILITY:
Inclusion Criteria:

* The specimen is a NPS or NS from a patient collected and preserved in 3 mL Universal Transport Media (UTM), BD Universal Viral Transport (UVT), or MicroTest M4RT transport media, or 1 mL Copan Eswab (Liquid Amies).
* The specimen is from a patient who is either hospitalized, admitted to a hospital emergency department, visiting an outpatient clinic or resident of a long-term care facility.
* The specimen is from a human patient with active signs and symptoms of respiratory tract infection at time of collection
* Specimen stored at 2-8°C for up to 72 hours from collection. If there is a delay in testing, store specimen at ≤-70 °C.
* The total volume of the leftover specimen received is ≥1.5 mL, except for specimens collected in Liquid Amies which requires a total leftover volume of ≥0.5 mL
* The specimen was received in good condition (no leakage or drying of the specimen).

Exclusion Criteria:

* Incorrect swab type
* Incorrect transport media
* Incorrect specimen handling (e.g. specimens not stored at recommended temperature)
* The specimen has undergone more than two freeze/thaw cycles
* Specimens collected with calcium alginate or organic swabs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy | Samples will be tested on LIAISON NES within two hours of collection.
  Estimates of Sensitivity/percent positive agreement (PPA) and Specificity/percent negative agreement (NPA) will be calculated based on a two-by-two table (comparator method result vs. result from LIAISON® NES FLU A/B, RSV & COVID-19 assay or LIAISON PLEX® RSP Flex assay) for each target. In addition, 95% two-sided confidence intervals will be provided. A separate Sensitivity/PPA and Specificity/NPA for each target, to include those specimens excluded due to a discrepancy between the standard-of-care and molecular comparator result, will be presented in a separate 2 x 2 table.

SECONDARY OUTCOMES:
Clinical Performance | Samples will be tested on LIAISON NES within one hour of collection.
  The secondary objective is to compare the clinical performance of the LIAISON NES FLU A/B, RSV & COVID-19 assay per clinical site, target patient sub-population (e.g. age group, patient location) and specimen collection method (e.g. professionally collected, patient self-collected).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - PAS Research - Henderson, Henderson, Nevada
  - PAS Research - Pittsburgh, Pittsburgh, Pennsylvania
  - PAS Research - McAllen, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No